CLINICAL TRIAL: NCT05427760
Title: Effect of Using Oxygen on the Diaper Dermatitis in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 386964
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-09

CONDITIONS: Diaper Rash; Diaper Dermatitis
Keywords: infant; diaper dermatitis; diaper rash; oxygen
MeSH Terms: conditions — Diaper Rash | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen Group (Experimental): After the baby's diaper is changed, an oxygen hose placed inside the diaper will provide free oxygen flow to the diaper area.
  Oxygen will be applied for 1 hour at each diaper change at a flow rate of 5L/min and at a concentration of 21% FiO2 which is equivalent to room air.
  Interventions: Drug: Oxygen
- Control Group (No Intervention): This group will only receive routine care: Diaper will be changed using disposable wet wipes and disposable baby diaper.
  A barrier cream containing 40% zinc oxide will be applied to the cleaned diaper area as a thin layer to cover the skin.
  Baby's diaper change will be done 8 times a day, every three hours.

INTERVENTIONS:
Drug: Oxygen — After changing the diaper, free flow oxygen will be provided to the diaper area for 1 hour with an oxygen cannula placed inside the diaper (oxygen flow is %21 Fio2, 5 L/min)
  Arms: Oxygen Group

SUMMARY:
Background: Airing the diaper area has a positive effect on dermatitis. In addition, it is reported in the literature that oxygen is effective in wound care. The aim of our study is to investigate the effect of oxygen on infant diaper dermatitis.

Method: The study population consisted of infants will admit to the neonatal intensive care unit of a public hospital in Istanbul between October 2022 and April 2023. Sixty newborns who met the study criteria will randomly divide into two as the experimental (n=30) and control (n=30) groups. Personal data form and diaper dermatitis observation form will be used to obtain the data. All babies' diapers will be changed 8 times a day. Oxygen flow will be applied to the experimental group for one hour after each diaper change. The degree of diaper dermatitis will be evaluated every 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Approved by the family for the study
* Born between 34-42. gestational weeks
* No skin disease other than diaper dermatitis
* No skin lesions of another disease other than dermatitis-related lesions in the gland area
* Newborns who has stable vital signs

Exclusion Criteria:

* Having a skin disease other than diaper dermatitis
* Having a lesion on the skin due to another disease
* Having a known skin allergy
* Born before 34. gestational weeks
* Having a gastrointestinal disease

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Diaper dermatitis healing scale result | 72 hours
  Expecting to healing diaper dermatitis symptoms at the time of intervention. The scale maximum value: 6 and minimum value: 0. As the scale score increases, the severity of dermatitis increases.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Dogan, Principal Investigator — Researcher Assistant
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abels C, Angelova-Fischer I. Skin Care Products: Age-Appropriate Cosmetics. Curr Probl Dermatol. 2018;54:173-182. doi: 10.1159/000489531. Epub 2018 Aug 21. PMID 30130785
- [Background] Ahmed B, Solanki B, Zaidi A, Khan MS, Musarrat J. Bacterial toxicity of biomimetic green zinc oxide nanoantibiotic: insights into ZnONP uptake and nanocolloid-bacteria interface. Toxicol Res (Camb). 2018 Dec 26;8(2):246-261. doi: 10.1039/c8tx00267c. eCollection 2019 Mar 1. PMID 30997024
- [Background] Almoudi MM, Hussein AS, Abu Hassan MI, Mohamad Zain N. A systematic review on antibacterial activity of zinc against Streptococcus mutans. Saudi Dent J. 2018 Oct;30(4):283-291. doi: 10.1016/j.sdentj.2018.06.003. Epub 2018 Jun 18. PMID 30202164
- [Background] Amer M, Diab N, Soliman M, Amer A. Neonatal skin care: what should we do? A four-week follow-up randomized controlled trial at Zagazig University Hospitals. Int J Dermatol. 2017 Nov;56(11):1198-1203. doi: 10.1111/ijd.13735. Epub 2017 Sep 7. PMID 28884798
- [Background] Atherton DJ. Understanding irritant napkin dermatitis. Int J Dermatol. 2016 Jul;55 Suppl 1:7-9. doi: 10.1111/ijd.13334. PMID 27311779
- [Background] Baurecht H, Ruhlemann MC, Rodriguez E, Thielking F, Harder I, Erkens AS, Stolzl D, Ellinghaus E, Hotze M, Lieb W, Wang S, Heinsen-Groth FA, Franke A, Weidinger S. Epidermal lipid composition, barrier integrity, and eczematous inflammation are associated with skin microbiome configuration. J Allergy Clin Immunol. 2018 May;141(5):1668-1676.e16. doi: 10.1016/j.jaci.2018.01.019. Epub 2018 Feb 5. PMID 29421277
- [Background] Bender JK, Faergemann J, Skold M. Skin Health Connected to the Use of Absorbent Hygiene Products: A Review. Dermatol Ther (Heidelb). 2017 Sep;7(3):319-330. doi: 10.1007/s13555-017-0189-y. Epub 2017 Jun 30. PMID 28667496
- [Background] Bennardo L, Del Duca E, Dastoli S, Schipani G, Scali E, Silvestri M, Nistico SP. Potential applications of topical oxygen therapy in dermatology. Dermatol Pract Concept. 2018 Oct 31;8(4):272-276. doi: 10.5826/dpc.0804a04. eCollection 2018 Oct. PMID 30479854
- [Background] Blume-Peytavi U, Kanti V. Prevention and treatment of diaper dermatitis. Pediatr Dermatol. 2018 Mar;35 Suppl 1:s19-s23. doi: 10.1111/pde.13495. PMID 29596731
- [Background] Blume-Peytavi U, Hauser M, Lunnemann L, Stamatas GN, Kottner J, Garcia Bartels N. Prevention of diaper dermatitis in infants--a literature review. Pediatr Dermatol. 2014 Jul-Aug;31(4):413-29. doi: 10.1111/pde.12348. Epub 2014 May 29. PMID 24890321
- [Background] Blume-Peytavi U, Lavender T, Jenerowicz D, Ryumina I, Stalder JF, Torrelo A, Cork MJ. Recommendations from a European Roundtable Meeting on Best Practice Healthy Infant Skin Care. Pediatr Dermatol. 2016 May;33(3):311-21. doi: 10.1111/pde.12819. Epub 2016 Feb 26. PMID 26919683
- [Background] Bonifaz A, Rojas R, Tirado-Sanchez A, Chavez-Lopez D, Mena C, Calderon L, Maria PO. Superficial Mycoses Associated with Diaper Dermatitis. Mycopathologia. 2016 Oct;181(9-10):671-9. doi: 10.1007/s11046-016-0020-9. Epub 2016 May 19. PMID 27193417
- [Background] Burdall O, Willgress L, Goad N. Neonatal skin care: Developments in care to maintain neonatal barrier function and prevention of diaper dermatitis. Pediatr Dermatol. 2019 Jan;36(1):31-35. doi: 10.1111/pde.13714. Epub 2018 Dec 2. PMID 30506880
- [Background] Caglar S, Yildiz GK, Bakoglu I, Salihoglu O. The Effect of Sunflower Seed and Almond Oil on Preterm Infant Skin: A Randomized Controlled Trial. Adv Skin Wound Care. 2020 Aug;33(8):1-6. doi: 10.1097/01.ASW.0000672500.18525.2e. PMID 32697476
- [Background] Carr AN, DeWitt T, Cork MJ, Eichenfield LF, Folster-Holst R, Hohl D, Lane AT, Paller A, Pickering L, Taieb A, Cui TY, Xu ZG, Wang X, Brink S, Niu Y, Ogle J, Odio M, Gibb RD. Diaper dermatitis prevalence and severity: Global perspective on the impact of caregiver behavior. Pediatr Dermatol. 2020 Jan;37(1):130-136. doi: 10.1111/pde.14047. Epub 2019 Dec 2. PMID 31793090
- [Background] Celeiro M, Lamas JP, Garcia-Jares C, Llompart M. Pressurized liquid extraction-gas chromatography-mass spectrometry analysis of fragrance allergens, musks, phthalates and preservatives in baby wipes. J Chromatogr A. 2015 Mar 6;1384:9-21. doi: 10.1016/j.chroma.2015.01.049. Epub 2015 Jan 22. PMID 25662066
- [Background] Chiabi A, Ngamgo Kamdem JC, Nkoro AG, Siyou H, Hamo S, Nguefack FD, Mah E, Nguefack S, Angwafo F 3rd. [Diaper rash and associated risk factors in infants at the Yaounde Gynaeco-obstetric and Pediatric Hospital, Cameroon]. Ann Dermatol Venereol. 2019 Feb;146(2):141-142. doi: 10.1016/j.annder.2018.07.017. Epub 2018 Dec 7. No abstract available. French. PMID 30527958
- [Background] Chiang N, Rodda OA, Sleigh J, Vasudevan T. Effects of topical negative pressure therapy on tissue oxygenation and wound healing in vascular foot wounds. J Vasc Surg. 2017 Aug;66(2):564-571. doi: 10.1016/j.jvs.2017.02.050. Epub 2017 Jun 2. PMID 28583732
- [Background] Chu DM, Ma J, Prince AL, Antony KM, Seferovic MD, Aagaard KM. Maturation of the infant microbiome community structure and function across multiple body sites and in relation to mode of delivery. Nat Med. 2017 Mar;23(3):314-326. doi: 10.1038/nm.4272. Epub 2017 Jan 23. PMID 28112736
- [Background] Cohen B. Differential Diagnosis of Diaper Dermatitis. Clin Pediatr (Phila). 2017 May;56(5_suppl):16S-22S. doi: 10.1177/0009922817706982. PMID 28420251
- [Background] Cooke A, Cork MJ, Victor S, Campbell M, Danby S, Chittock J, Lavender T. Olive Oil, Sunflower Oil or no Oil for Baby Dry Skin or Massage: A Pilot, Assessor-blinded, Randomized Controlled Trial (the Oil in Baby SkincaRE [OBSeRvE] Study). Acta Derm Venereol. 2016 Mar;96(3):323-30. doi: 10.2340/00015555-2279. PMID 26551528
- [Background] Cooke A, Bedwell C, Campbell M, McGowan L, Ersser SJ, Lavender T. Skin care for healthy babies at term: A systematic review of the evidence. Midwifery. 2018 Jan;56:29-43. doi: 10.1016/j.midw.2017.10.001. Epub 2017 Oct 6. PMID 29055852
- [Background] Coughlin CC, Eichenfield LF, Frieden IJ. Diaper dermatitis: clinical characteristics and differential diagnosis. Pediatr Dermatol. 2014 Nov;31 Suppl 1:19-24. doi: 10.1111/pde.12500. PMID 25403935
- [Background] Counts J, Weisbrod A, Yin S. Common Diaper Ingredient Questions: Modern Disposable Diaper Materials Are Safe and Extensively Tested. Clin Pediatr (Phila). 2017 May;56(5_suppl):23S-27S. doi: 10.1177/0009922817706998. PMID 28420254
- [Background] Cundell AM. Microbial Ecology of the Human Skin. Microb Ecol. 2018 Jul;76(1):113-120. doi: 10.1007/s00248-016-0789-6. Epub 2016 May 31. PMID 27245597
- [Background] Dey S, Helmes CT, White JC, Zhou S. Safety of Disposable Diaper Materials: Extensive Evaluations Validate Use. Clin Pediatr (Phila). 2014 Aug;53(9 suppl):17S-19S. doi: 10.1177/0009922814540378. Epub 2014 Jun 24. PMID 24961774
- [Background] Dall'Oglio F, Musumeci ML, Puglisi DF, Micali G. A novel treatment of diaper dermatitis in children and adults. J Cosmet Dermatol. 2021 Apr;20 Suppl 1(Suppl 1):1-4. doi: 10.1111/jocd.14091. PMID 33934478
- [Background] Dey S, Kenneally D, Odio M, Hatzopoulos I. Modern diaper performance: construction, materials, and safety review. Int J Dermatol. 2016 Jul;55 Suppl 1:18-20. doi: 10.1111/ijd.13333. PMID 27311782
- [Background] Dimitriu PA, Iker B, Malik K, Leung H, Mohn WW, Hillebrand GG. New Insights into the Intrinsic and Extrinsic Factors That Shape the Human Skin Microbiome. mBio. 2019 Jul 2;10(4):e00839-19. doi: 10.1128/mBio.00839-19. PMID 31266865
- [Background] Kozic Dokmanovic S, Kolovrat K, Laskaj R, Jukic V, Vrkic N, Begovac J. Effect of Extra Virgin Olive Oil on Biomarkers of Inflammation in HIV-Infected Patients: A Randomized, Crossover, Controlled Clinical Trial. Med Sci Monit. 2015 Aug 16;21:2406-13. doi: 10.12659/MSM.893881. PMID 26280823
- [Background] El-Ashram S, El-Samad LM, Basha AA, El Wakil A. Naturally-derived targeted therapy for wound healing: Beyond classical strategies. Pharmacol Res. 2021 Aug;170:105749. doi: 10.1016/j.phrs.2021.105749. Epub 2021 Jun 30. PMID 34214630
- [Background] Elias PM. The how, why and clinical importance of stratum corneum acidification. Exp Dermatol. 2017 Nov;26(11):999-1003. doi: 10.1111/exd.13329. Epub 2017 May 12. PMID 28266738
- [Background] Ersoy-Evans S, Akinci H, Dogan S, Atakan N. Diaper Dermatitis: A Review of 63 Children. Pediatr Dermatol. 2016 May;33(3):332-6. doi: 10.1111/pde.12860. Epub 2016 Apr 4. PMID 27040137
- [Background] Esser MS, Johnson TS. An Integrative Review of Clinical Characteristics of Infants With Diaper Dermatitis. Adv Neonatal Care. 2020 Aug;20(4):276-285. doi: 10.1097/ANC.0000000000000682. PMID 31895136
- [Background] Esser M. Diaper Dermatitis: What Do We Do Next? Adv Neonatal Care. 2016 Oct;16 Suppl 5S:S21-S25. doi: 10.1097/ANC.0000000000000316. PMID 27676110
- [Background] Felter SP, Carr AN, Zhu T, Kirsch T, Niu G. Safety evaluation for ingredients used in baby care products: Consideration of diaper rash. Regul Toxicol Pharmacol. 2017 Nov;90:214-221. doi: 10.1016/j.yrtph.2017.09.011. Epub 2017 Sep 12. PMID 28916467
- [Background] Fluhr JW, Darlenski R. Skin Surface pH in Newborns: Origin and Consequences. Curr Probl Dermatol. 2018;54:26-32. doi: 10.1159/000489515. Epub 2018 Aug 21. PMID 30130770
- [Background] Folster-Holst R, Sunderkotter C. [Scabies in childhood and adolescence]. Hautarzt. 2016 Dec;67(12):1007-1020. doi: 10.1007/s00105-016-3901-4. German. PMID 27826663
- [Background] Folster-Holst R. Differential diagnoses of diaper dermatitis. Pediatr Dermatol. 2018 Mar;35 Suppl 1:s10-s18. doi: 10.1111/pde.13484. PMID 29596730
- [Background] Frykberg RG. Topical Wound Oxygen Therapy in the Treatment of Chronic Diabetic Foot Ulcers. Medicina (Kaunas). 2021 Aug 31;57(9):917. doi: 10.3390/medicina57090917. PMID 34577840
- [Background] Gottrup F, Dissemond J, Baines C, Frykberg R, Jensen PO, Kot J, Kroger K, Longobardi P. Use of Oxygen Therapies in Wound Healing. J Wound Care. 2017 May 1;26(Sup5):S1-S43. doi: 10.12968/jowc.2017.26.Sup5.S1. No abstract available. PMID 28475468
- [Background] Gustin J, Gibb R, Maltbie D, Roe D, Waimin Siu S. The impact of diaper design on mitigating known causes of diaper dermatitis. Pediatr Dermatol. 2018 Nov;35(6):792-795. doi: 10.1111/pde.13680. Epub 2018 Aug 30. PMID 30168199
- [Background] Gustin J, Bohman L, Ogle J, Chaudhary T, Li L, Fadayel G, Mitchell MC, Narendran V, Visscher MO, Carr AN. Use of an emollient-containing diaper and pH-buffered wipe regimen restores skin pH and reduces residual enzymatic activity. Pediatr Dermatol. 2020 Jul;37(4):626-631. doi: 10.1111/pde.14169. Epub 2020 Apr 21. PMID 32314466
- [Background] Gustin J, Bohman L, Ogle J, Fadayel G, Mitchell MC, Narendran V, Visscher MO, Carr AN. Improving newborn skin health: Effects of diaper care regimens on skin pH and erythema. Pediatr Dermatol. 2021 Jul;38(4):768-774. doi: 10.1111/pde.14602. Epub 2021 May 31. PMID 34060142
- [Background] Haller HL, Sander F, Popp D, Rapp M, Hartmann B, Demircan M, Nischwitz SP, Kamolz LP. Oxygen, pH, Lactate, and Metabolism-How Old Knowledge and New Insights Might Be Combined for New Wound Treatment. Medicina (Kaunas). 2021 Nov 1;57(11):1190. doi: 10.3390/medicina57111190. PMID 34833408
- [Background] Hayes PD, Alzuhir N, Curran G, Loftus IM. Topical oxygen therapy promotes the healing of chronic diabetic foot ulcers: a pilot study. J Wound Care. 2017 Nov 2;26(11):652-660. doi: 10.12968/jowc.2017.26.11.652. PMID 29131746
- [Background] Hebert AA. A new therapeutic horizon in diaper dermatitis: Novel agents with novel action. Int J Womens Dermatol. 2021 Feb 16;7(4):466-470. doi: 10.1016/j.ijwd.2021.02.003. eCollection 2021 Sep. PMID 34621960
- [Background] Jeong E, Kim CU, Byun J, Lee J, Kim HE, Kim EJ, Choi KJ, Hong SW. Quantitative evaluation of the antibacterial factors of ZnO nanorod arrays under dark conditions: Physical and chemical effects on Escherichia coli inactivation. Sci Total Environ. 2020 Apr 10;712:136574. doi: 10.1016/j.scitotenv.2020.136574. Epub 2020 Jan 8. PMID 32050388
- [Background] Johnson E, Hunt R. Infant skin care: updates and recommendations. Curr Opin Pediatr. 2019 Aug;31(4):476-481. doi: 10.1097/MOP.0000000000000791. PMID 31188166
- [Background] Johnson DE. Extremely Preterm Infant Skin Care: A Transformation of Practice Aimed to Prevent Harm. Adv Neonatal Care. 2016 Oct;16 Suppl 5S:S26-S32. doi: 10.1097/ANC.0000000000000335. PMID 27676111
- [Background] Kanti V, Gunther M, Stroux A, Sawatzky S, Henrich W, Abou-Dakn M, Blume-Peytavi U, Garcia Bartels N. Influence of sunflower seed oil or baby lotion on the skin barrier function of newborns: A pilot study. J Cosmet Dermatol. 2017 Dec;16(4):500-507. doi: 10.1111/jocd.12302. Epub 2017 Jan 10. PMID 28070970
- [Background] Kaufman H, Gurevich M, Tamir E, Keren E, Alexander L, Hayes P. Topical oxygen therapy stimulates healing in difficult, chronic wounds: a tertiary centre experience. J Wound Care. 2018 Jul 2;27(7):426-433. doi: 10.12968/jowc.2018.27.7.426. PMID 30016136
- [Background] Keshavarz A, Zeinaloo AA, Mahram M, Mohammadi N, Sadeghpour O, Maleki MR. Efficacy of Traditional Medicine Product Henna and Hydrocortisone on Diaper Dermatitis in Infants. Iran Red Crescent Med J. 2016 Feb 22;18(5):e24809. doi: 10.5812/ircmj.24809. eCollection 2016 May. PMID 27478628
- [Background] Khalifian S, Golden WC, Cohen BA. Skin care practices in newborn nurseries and mother-baby units in Maryland. J Perinatol. 2017 Jun;37(6):615-621. doi: 10.1038/jp.2016.226. Epub 2016 Dec 22. PMID 28005064
- [Background] Kirchner F, Capone KA, Mack MC, Stamatas GN. Expression of cutaneous immunity markers during infant skin maturation. Pediatr Dermatol. 2018 Jul;35(4):468-471. doi: 10.1111/pde.13516. Epub 2018 Apr 25. PMID 29691908
- [Background] Klunk C, Domingues E, Wiss K. An update on diaper dermatitis. Clin Dermatol. 2014 Jul-Aug;32(4):477-87. doi: 10.1016/j.clindermatol.2014.02.003. Epub 2014 Feb 28. PMID 25017459
- [Background] Kuller JM. Infant Skin Care Products: What Are the Issues? Adv Neonatal Care. 2016 Oct;16 Suppl 5S:S3-S12. doi: 10.1097/ANC.0000000000000341. PMID 27676112
- [Background] Kusari A, Han AM, Virgen CA, Matiz C, Rasmussen M, Friedlander SF, Eichenfield DZ. Evidence-based skin care in preterm infants. Pediatr Dermatol. 2019 Jan;36(1):16-23. doi: 10.1111/pde.13725. Epub 2018 Dec 12. PMID 30548578
- [Background] Li Y, Liao C, Tjong SC. Recent Advances in Zinc Oxide Nanostructures with Antimicrobial Activities. Int J Mol Sci. 2020 Nov 22;21(22):8836. doi: 10.3390/ijms21228836. PMID 33266476
- [Background] Lim YSL, Carville K. Prevention and Management of Incontinence-Associated Dermatitis in the Pediatric Population: An Integrative Review. J Wound Ostomy Continence Nurs. 2019 Jan/Feb;46(1):30-37. doi: 10.1097/WON.0000000000000490. PMID 30608338
- [Background] Liou YL, Ericson ME, Warshaw EM. Formaldehyde Release From Baby Wipes: Analysis Using the Chromotropic Acid Method. Dermatitis. 2019 May/Jun;30(3):207-212. doi: 10.1097/DER.0000000000000478. PMID 31045936
- [Background] Liu Q, Zhang Y, Danby SG, Cork MJ, Stamatas GN. Infant Skin Barrier, Structure, and Enzymatic Activity Differ from Those of Adult in an East Asian Cohort. Biomed Res Int. 2018 Jul 12;2018:1302465. doi: 10.1155/2018/1302465. eCollection 2018. PMID 30112358
- [Background] Lu J, Li M, Huang J, Gao L, Pan Y, Fu Z, Dou J, Huang J, Xiang Y. [Effect of ozone on Staphylococcus aureus colonization in patients with atopic dermatitis]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2018 Feb 28;43(2):157-162. doi: 10.11817/j.issn.1672-7347.2018.02.009. Chinese. PMID 29559599
- [Background] Ludriksone L, Garcia Bartels N, Kanti V, Blume-Peytavi U, Kottner J. Skin barrier function in infancy: a systematic review. Arch Dermatol Res. 2014 Sep;306(7):591-9. doi: 10.1007/s00403-014-1458-6. Epub 2014 Mar 5. PMID 24595645
- [Background] Lukowski AF, Liu X, Peirano P, Odio M, Bauer PJ. Disposable diaper use promotes consolidated nighttime sleep and positive mother-infant interactions in Chinese 6-month-olds. J Fam Psychol. 2015 Jun;29(3):371-81. doi: 10.1037/fam0000072. Epub 2015 May 4. PMID 25938711
- [Background] Mactaggart E, Orchard D, Mui Tam M. Baby wipes and nappy rash - what is the relationship? A review. Australas J Dermatol. 2021 Nov;62(4):470-477. doi: 10.1111/ajd.13715. Epub 2021 Sep 15. PMID 34523734
- [Background] Mahmoudi M, Adib-Hajbaghery M, Mashaiekhi M. Comparing the effects of Bentonite & Calendula on the improvement of infantile diaper dermatitis: A randomized controlled trial. Indian J Med Res. 2015 Dec;142(6):742-6. doi: 10.4103/0971-5916.174567. PMID 26831423
- [Background] Malik A, Witsberger E, Cottrell L, Kiefer A, Yossuck P. Perianal Dermatitis, Its Incidence, and Patterns of Topical Therapies in a Level IV Neonatal Intensive Care Unit. Am J Perinatol. 2018 Apr;35(5):486-493. doi: 10.1055/s-0037-1608708. Epub 2017 Nov 22. PMID 29166675
- [Background] Merrill L. Prevention, Treatment and Parent Education for Diaper Dermatitis. Nurs Womens Health. 2015 Aug-Sep;19(4):324-36; quiz 337. doi: 10.1111/1751-486X.12218. PMID 26264797
- [Background] Mews J, Tomaszewska A, Siewiera J, Lewicki S, Kuczborska K, Lipinska-Opalka A, Kalicki B. Effects of Hyperbaric Oxygen Therapy in Children with Severe Atopic Dermatitis. J Clin Med. 2021 Mar 10;10(6):1157. doi: 10.3390/jcm10061157. PMID 33802050
- [Background] Mooney E, Rademaker M, Dailey R, Daniel BS, Drummond C, Fischer G, Foster R, Grills C, Halbert A, Hill S, King E, Leins E, Morgan V, Phillips RJ, Relic J, Rodrigues M, Scardamaglia L, Smith S, Su J, Wargon O, Orchard D. Adverse effects of topical corticosteroids in paediatric eczema: Australasian consensus statement. Australas J Dermatol. 2015 Nov;56(4):241-51. doi: 10.1111/ajd.12313. Epub 2015 Mar 6. PMID 25752907
- [Background] Mota AC, de Castro RD, de Araujo Oliveira J, de Oliveira Lima E. Antifungal Activity of Apple Cider Vinegar on Candida Species Involved in Denture Stomatitis. J Prosthodont. 2015 Jun;24(4):296-302. doi: 10.1111/jopr.12207. Epub 2014 Sep 14. PMID 25219289
- [Background] Nataraj M, Maiya AG, Karkada G, Hande M, Rodrigues GS, Shenoy R, Prasad SS. Application of Topical Oxygen Therapy in Healing Dynamics of Diabetic Foot Ulcers - A Systematic Review. Rev Diabet Stud. 2019;15:74-82. doi: 10.1900/RDS.2019.15.74. Epub 2019 Dec 30. PMID 31904759
- [Background] Niederauer MQ. How can we deliver oxygen to wounds? J Wound Care. 2021 May 1;30(Sup5):S3-S4. doi: 10.12968/jowc.2021.30.Sup5.S3. No abstract available. PMID 33979233
- [Background] Nourbakhsh SM, Rouhi-Boroujeni H, Kheiri M, Mobasheri M, Shirani M, Ahrani S, Karami J, Hafshejani ZK. Effect of Topical Application of the Cream Containing Magnesium 2% on Treatment of Diaper Dermatitis and Diaper Rash in Children A Clinical Trial Study. J Clin Diagn Res. 2016 Jan;10(1):WC04-6. doi: 10.7860/JCDR/2016/14997.7143. Epub 2016 Jan 1. PMID 26894161
- [Background] O'Connor RJ, Sanchez V, Wang Y, Gibb R, Nofziger DL, Bailey M, Carr AN. Evaluation of the Impact of 2 Disposable Diapers in the "Natural" Diaper Category on Diapered Skin Condition. Clin Pediatr (Phila). 2019 Jun;58(7):806-815. doi: 10.1177/0009922819841136. Epub 2019 Apr 9. PMID 30961367
- [Background] Oranje AP, de Waard-van der Spek FB. Recent developments in the management of common childhood skin infections. J Infect. 2015 Jun;71 Suppl 1:S76-9. doi: 10.1016/j.jinf.2015.04.030. Epub 2015 Apr 29. PMID 25936745
- [Background] Ozdemir A, Bas VN. Iatrogenic Cushing's syndrome due to overuse of topical steroid in the diaper area. J Trop Pediatr. 2014 Oct;60(5):404-6. doi: 10.1093/tropej/fmu036. Epub 2014 Jul 11. No abstract available. PMID 25016382
- [Background] Pammi M, O'Brien JL, Ajami NJ, Wong MC, Versalovic J, Petrosino JF. Development of the cutaneous microbiome in the preterm infant: A prospective longitudinal study. PLoS One. 2017 Apr 27;12(4):e0176669. doi: 10.1371/journal.pone.0176669. eCollection 2017. PMID 28448623
- [Background] Patrizi A, Neri I, Ricci G, Cipriani F, Ravaioli GM. Advances in pharmacotherapeutic management of common skin diseases in neonates and infants. Expert Opin Pharmacother. 2017 May;18(7):717-725. doi: 10.1080/14656566.2017.1316371. Epub 2017 Apr 21. PMID 28429969
- [Background] Hertis Petek T, Petek M, Petek T, Marcun Varda N. Emerging Links between Microbiome Composition and Skin Immunology in Diaper Dermatitis: A Narrative Review. Children (Basel). 2022 Jan 15;9(1):112. doi: 10.3390/children9010112. PMID 35053737
- [Background] Sikic Pogacar M, Maver U, Marcun Varda N, Micetic-Turk D. Diagnosis and management of diaper dermatitis in infants with emphasis on skin microbiota in the diaper area. Int J Dermatol. 2018 Mar;57(3):265-275. doi: 10.1111/ijd.13748. Epub 2017 Oct 6. PMID 28986935
- [Background] Proksch E, de Bony R, Trapp S, Boudon S. Topical use of dexpanthenol: a 70th anniversary article. J Dermatolog Treat. 2017 Dec;28(8):766-773. doi: 10.1080/09546634.2017.1325310. Epub 2017 May 14. PMID 28503966
- [Background] Rao C, Xiao L, Liu H, Li S, Lu J, Li J, Gu S. Effects of topical oxygen therapy on ischemic wound healing. J Phys Ther Sci. 2016 Jan;28(1):118-23. doi: 10.1589/jpts.28.118. Epub 2016 Jan 30. PMID 26957741
- [Background] Rippke F, Berardesca E, Weber TM. pH and Microbial Infections. Curr Probl Dermatol. 2018;54:87-94. doi: 10.1159/000489522. Epub 2018 Aug 21. PMID 30130777
- [Background] Sechi LA, Melis A, Pala A, Marigliano A, Sechi G, Tedde R. Serum insulin, insulin sensitivity, and erythrocyte sodium metabolism in normotensive and essential hypertensive subjects with and without overweight. Clin Exp Hypertens A. 1991;13(2):261-76. doi: 10.3109/10641969109042062. PMID 2065466
- [Background] Rogers S, Thomas M, Chan B, Hinckley SK, Henderson C. A Quality Improvement Approach to Perineal Skin Care: Using Standardized Guidelines and Novel Diaper Wipes to Reduce Diaper Dermatitis in NICU Infants. Adv Neonatal Care. 2021 Jun 1;21(3):189-197. doi: 10.1097/ANC.0000000000000795. PMID 33009153
- [Background] Sarkar R, Podder I, Gokhale N, Jagadeesan S, Garg VK. Use of vegetable oils in dermatology: an overview. Int J Dermatol. 2017 Nov;56(11):1080-1086. doi: 10.1111/ijd.13623. Epub 2017 Apr 19. PMID 28421610
- [Background] Schneider AM, Nelson AM. Skin microbiota: Friend or foe in pediatric skin health and skin disease. Pediatr Dermatol. 2019 Nov;36(6):815-822. doi: 10.1111/pde.13955. Epub 2019 Oct 6. PMID 31588632
- [Background] Seifi B, Jalali S, Heidari M. Assessment Effect of Breast Milk on Diaper Dermatitis. Dermatol Reports. 2017 Mar 13;9(1):7044. doi: 10.4081/dr.2017.7044. eCollection 2017 Mar 13. PMID 28626535
- [Background] Serena TE, Bullock NM, Cole W, Lantis J, Li L, Moore S, Patel K, Sabo M, Wahab N, Price P. Topical oxygen therapy in the treatment of diabetic foot ulcers: a multicentre, open, randomised controlled clinical trial. J Wound Care. 2021 May 1;30(Sup5):S7-S14. doi: 10.12968/jowc.2021.30.Sup5.S7. PMID 33979229
- [Background] Shane AL, Sanchez PJ, Stoll BJ. Neonatal sepsis. Lancet. 2017 Oct 14;390(10104):1770-1780. doi: 10.1016/S0140-6736(17)31002-4. Epub 2017 Apr 20. PMID 28434651
- [Background] Sharifi-Heris Z, Farahani LA, Haghani H, Abdoli-Oskouee S, Hasanpoor-Azghady SB. Comparison the effects of topical application of olive and calendula ointments on Children's diaper dermatitis: A triple-blind randomized clinical trial. Dermatol Ther. 2018 Nov;31(6):e12731. doi: 10.1111/dth.12731. Epub 2018 Oct 12. PMID 30311724
- [Background] Simonetti O, Bacchetti T, Ferretti G, Molinelli E, Rizzetto G, Bellachioma L, Offidani A. Oxidative Stress and Alterations of Paraoxonases in Atopic Dermatitis. Antioxidants (Basel). 2021 Apr 28;10(5):697. doi: 10.3390/antiox10050697. PMID 33925093
- [Background] Singh A, Panda K, Mishra J, Dash A. A Comparative Study between Indigenous Low Cost Negative Pressure Wound Therapy with Added Local Oxygen versus Conventional Negative Pressure Wound Therapy. Malays Orthop J. 2020 Nov;14(3):129-136. doi: 10.5704/MOJ.2011.020. PMID 33403073
- [Background] de Smet GHJ, Kroese LF, Menon AG, Jeekel J, van Pelt AWJ, Kleinrensink GJ, Lange JF. Oxygen therapies and their effects on wound healing. Wound Repair Regen. 2017 Aug;25(4):591-608. doi: 10.1111/wrr.12561. Epub 2017 Aug 7. PMID 28783878
- [Background] Song Z, Guo X, Zhang X. Effects of topical oxygen therapy on chronic traumatic wounds and its impact on granulation tissue. Am J Transl Res. 2021 Jun 15;13(6):7294-7299. eCollection 2021. PMID 34306496
- [Background] Stamatas GN, Tierney NK. Diaper dermatitis: etiology, manifestations, prevention, and management. Pediatr Dermatol. 2014 Jan-Feb;31(1):1-7. doi: 10.1111/pde.12245. Epub 2013 Nov 14. PMID 24224482
- [Background] Stamatas GN, Bensaci J, Greugny E, Kaur S, Wang H, Dizon MV, Cork MJ, Friedman AJ, Oddos T. A Predictive Self-Organizing Multicellular Computational Model of Infant Skin Permeability to Topically Applied Substances. J Invest Dermatol. 2021 Aug;141(8):2049-2055.e1. doi: 10.1016/j.jid.2021.02.012. Epub 2021 Mar 9. PMID 33705796
- [Background] Stewart D, Benitz W; COMMITTEE ON FETUS AND NEWBORN. Umbilical Cord Care in the Newborn Infant. Pediatrics. 2016 Sep;138(3):e20162149. doi: 10.1542/peds.2016-2149. PMID 27573092
- [Background] Sukhneewat C, Chaiyarit J, Techasatian L. Diaper dermatitis: a survey of risk factors in Thai children aged under 24 months. BMC Dermatol. 2019 Jul 2;19(1):7. doi: 10.1186/s12895-019-0089-1. PMID 31262288
- [Background] Taieb A. Skin barrier in the neonate. Pediatr Dermatol. 2018 Mar;35 Suppl 1:s5-s9. doi: 10.1111/pde.13482. PMID 29596733
- [Background] Teufel A, Howard B, Hu P, Carr AN. Characterization of the microbiome in the infant diapered area: Insights from healthy and damaged skin. Exp Dermatol. 2021 Oct;30(10):1409-1417. doi: 10.1111/exd.14198. Epub 2020 Oct 13. PMID 32974911
- [Background] Thanigaimani S, Singh T, Golledge J. Topical oxygen therapy for diabetes-related foot ulcers: A systematic review and meta-analysis. Diabet Med. 2021 Aug;38(8):e14585. doi: 10.1111/dme.14585. Epub 2021 Apr 29. PMID 33871095
- [Background] Committee to Review the Formaldehyde Assessment in the National Toxicology Program 12th Report on Carcinogens; Board on Environmental Studies and Toxicology; Division on Earth and Life Sciences; National Research Council. Review of the Formaldehyde Assessment in the National Toxicology Program 12th Report on Carcinogens. Washington (DC): National Academies Press (US); 2014 Sep 8. Available from http://www.ncbi.nlm.nih.gov/books/NBK248276/ PMID 25340250
- [Background] Timm CM, Loomis K, Stone W, Mehoke T, Brensinger B, Pellicore M, Staniczenko PPA, Charles C, Nayak S, Karig DK. Isolation and characterization of diverse microbial representatives from the human skin microbiome. Microbiome. 2020 Apr 22;8(1):58. doi: 10.1186/s40168-020-00831-y. PMID 32321582
- [Background] Tuzun Y, Wolf R, Baglam S, Engin B. Diaper (napkin) dermatitis: A fold (intertriginous) dermatosis. Clin Dermatol. 2015 Jul-Aug;33(4):477-82. doi: 10.1016/j.clindermatol.2015.04.012. Epub 2015 Apr 9. PMID 26051065
- [Background] Underwood MA, Sohn K. The Microbiota of the Extremely Preterm Infant. Clin Perinatol. 2017 Jun;44(2):407-427. doi: 10.1016/j.clp.2017.01.005. Epub 2017 Mar 22. PMID 28477669
- [Background] Van Gysel D. Infections and skin diseases mimicking diaper dermatitis. Int J Dermatol. 2016 Jul;55 Suppl 1:10-3. doi: 10.1111/ijd.13372. PMID 27311780
- [Background] Visscher M, Narendran V. The Ontogeny of Skin. Adv Wound Care (New Rochelle). 2014 Apr 1;3(4):291-303. doi: 10.1089/wound.2013.0467. PMID 24761361
- [Background] Visscher MO, Adam R, Brink S, Odio M. Newborn infant skin: physiology, development, and care. Clin Dermatol. 2015 May-Jun;33(3):271-80. doi: 10.1016/j.clindermatol.2014.12.003. Epub 2014 Dec 8. PMID 25889127
- [Background] Visscher MO, Burkes SA, Adams DM, Hammill AM, Wickett RR. Infant skin maturation: Preliminary outcomes for color and biomechanical properties. Skin Res Technol. 2017 Nov;23(4):545-551. doi: 10.1111/srt.12369. Epub 2017 Mar 16. PMID 28303612
- [Background] Vongsa R, Rodriguez K, Koenig D, Cunningham C. Benefits of Using an Appropriately Formulated Wipe to Clean Diapered Skin of Preterm Infants. Glob Pediatr Health. 2019 Feb 19;6:2333794X19829186. doi: 10.1177/2333794X19829186. eCollection 2019. PMID 30815515
- [Background] Ward TL, Dominguez-Bello MG, Heisel T, Al-Ghalith G, Knights D, Gale CA. Development of the Human Mycobiome over the First Month of Life and across Body Sites. mSystems. 2018 Mar 6;3(3):e00140-17. doi: 10.1128/mSystems.00140-17. eCollection 2018 May-Jun. PMID 29546248
- [Background] Warshaw EM, Aschenbeck KA, Zug KA, Belsito DV, Zirwas MJ, Fowler JF Jr, Taylor JS, Sasseville D, Fransway AF, DeLeo VA, Marks JG Jr, Pratt MD, Maibach HI, Mathias CG, DeKoven JG. Wet Wipe Allergens: Retrospective Analysis From the North American Contact Dermatitis Group 2011-2014. Dermatitis. 2017 Jan/Feb;28(1):64-69. doi: 10.1097/DER.0000000000000248. PMID 28002231
- [Background] Weidinger S, Novak N. Atopic dermatitis. Lancet. 2016 Mar 12;387(10023):1109-1122. doi: 10.1016/S0140-6736(15)00149-X. Epub 2015 Sep 13. PMID 26377142
- [Background] Yip WL. Influence of oxygen on wound healing. Int Wound J. 2015 Dec;12(6):620-4. doi: 10.1111/iwj.12324. Epub 2014 Jun 26. PMID 24974913
- [Background] Yonezawa K, Haruna M, Matsuzaki M, Shiraishi M, Kojima R. Effects of moisturizing skincare on skin barrier function and the prevention of skin problems in 3-month-old infants: A randomized controlled trial. J Dermatol. 2018 Jan;45(1):24-30. doi: 10.1111/1346-8138.14080. Epub 2017 Oct 6. PMID 28983938
- [Background] Younge NE, Araujo-Perez F, Brandon D, Seed PC. Early-life skin microbiota in hospitalized preterm and full-term infants. Microbiome. 2018 May 31;6(1):98. doi: 10.1186/s40168-018-0486-4. PMID 29855335
- [Background] Yu J, Treat J, Chaney K, Brod B. Potential Allergens in Disposable Diaper Wipes, Topical Diaper Preparations, and Disposable Diapers: Under-recognized Etiology of Pediatric Perineal Dermatitis. Dermatitis. 2016 May-Jun;27(3):110-8. doi: 10.1097/DER.0000000000000177. PMID 27172304
- [Background] Yuan C, Takagi R, Yao XQ, Xu YF, Ishida K, Toyoshima H. Comparison of the Effectiveness of New Material Diapers versus Standard Diapers for the Prevention of Diaper Rash in Chinese Babies: A Double-Blinded, Randomized, Controlled, Cross-Over Study. Biomed Res Int. 2018 Jun 24;2018:5874184. doi: 10.1155/2018/5874184. eCollection 2018. PMID 30035123
- [Background] Zeng J, Dou J, Gao L, Xiang Y, Huang J, Ding S, Chen J, Zeng Q, Luo Z, Tan W, Lu J. Topical ozone therapy restores microbiome diversity in atopic dermatitis. Int Immunopharmacol. 2020 Mar;80:106191. doi: 10.1016/j.intimp.2020.106191. Epub 2020 Jan 24. PMID 31986325
- [Background] Zheng Y, Wang Q, Ma L, Chen Y, Gao Y, Zhang G, Cui S, Liang H, Song L, He C. Shifts in the skin microbiome associated with diaper dermatitis and emollient treatment amongst infants and toddlers in China. Exp Dermatol. 2019 Nov;28(11):1289-1297. doi: 10.1111/exd.14028. Epub 2019 Sep 16. PMID 31472099